CLINICAL TRIAL: NCT03881618
Title: the Efficacy of Electro-acupuncture Therapy for Patients With Methadone Maintenance Treatment : a Randomized Control Trial
Brief Title: Efficacy of Electro-Acupuncture Therapy for Patients With Methadone Maintenance Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Principal Investigator, Chung-Hua Hsu, Clinical Professor, Taipei City Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TCHIRB-10601106
Record Dates: First submitted 2018-10-02; First posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Sleep Disorder (Disorder)
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: two group . a group and b group. the intervention of a group is electroacupuncture + auricular pressure and b group is auricular pressure ,after intervention for 1 month and crossover.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electroacupuncture+auricular pressure (Experimental): a group :electroacupuncture+auricular pressure for 20 minutes twice a week for 4 weeks
  Interventions: Procedure: electroacupuncture+auricular pressure,
- auricular pressure (Active Comparator): b group :auricular pressure for 20 minutes twice a week for 4 weeks.
  Interventions: Procedure: electroacupuncture+auricular pressure,

INTERVENTIONS:
Procedure: electroacupuncture+auricular pressure, — electroacupuncture+auricular pressure for 20 minutes
  Other Names: auricular pressure

SUMMARY:
The population of drug abuse(heroin) had reached about 200,000 in Taiwan, and the age distribution is mainly in young adults. The social, medical and economic problems of drug addiction are profound and include lost productivity, disrupted relationships, crime and violence, HIV/AIDS and other infectious diseases. Methadone substitution therapy has been the treatment of first choice for opiate dependence, but patient on Methadone substitution therapy report a wide side effects, and relapse rate is up to two third of methadone treatment patients between one to two years.

This research is aim to build a development model. First of all, investigators plan to review some convincing articles and then analyze the efficacy of TCM in drug addiction. According to review articles and experience of professionals, investigators establish a model for TCM included in addiction treatment. Investigators will cooperate with Western medicine together , through common assessment scales to confirm the efficacy of traditional Chinese medicine and compare with current routine treatment.

DETAILED DESCRIPTION:
Drug addiction is a chronic medical illness and an important public health problem worldwide. The population of drug abuse had reached about 200,000 in Taiwan, and the age distribution is mainly in young adults. The social, medical and economic problems of drug addiction are profound and include lost productivity, disrupted relationships, crime and violence, HIV/AIDS and other infectious diseases. Therefore, drug addiction treatment is a hot issue of Ministry of Health and Welfare . Methadone substitution therapy has been the treatment of first choice for opiate dependence, but patient on Methadone substitution therapy report a wide side effects, and relapse rate is up to two third of methadone treatment patients between one to two years. Therefore, adjuvant therapeutic interventions for drug addiction patients are needed. Contrast to conventional Western medicine, traditional Chinese medicine is the most common used therapy of complementary and alternative medicine. However, traditional Chinese medicine (TCM) was excluded from the service for drug addiction treatment. Investigators need to establish a model for TCM as an alternative therapy included in addiction treatment and provide a better care system for drug addiction.

This research is aim to build a development model. First of all, investigators plan to review some convincing articles and then analyze the efficacy of TCM in drug addiction. According to review articles and experience of professionals, we establish a model for TCM included in addiction treatment. Investigators will cooperate with Western medicine together , through common assessment scales to confirm the efficacy of traditional Chinese medicine and compare with current routine treatment. According to above experience, investigators provide a Standard Operation Procedure for TCM treatment for drug addiction and policy suggestion. For drug addiction , this factually achieves communication and integration of Chinese and Western medicine, and benefits the public.

ELIGIBILITY:
Inclusion Criteria:

* Comply with Diagnostic Guidelines for Mental Disorders (DSM-V) for diagnosis of opioid use disorders
* Rules accepting Methadone Maintenance Therapy
* Patients between the ages of 20 and 65.

Exclusion Criteria:

* Unacceptable for research content.
* The detector cannot be completed.
* Unwilling to cooperate with acupuncture and ear beans.
* Those whose vital signs are unstable.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-04-21 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | 20 months
  The highest score in the whole questionnaire is 21 point, and the lowest score is 0 points.The lower the score, the better the sleep quality
Severity of Dependence Scale | 20 months
  The highest score in the whole questionnaire is 15 point, and the lowest score is 0 points. The higher the score, the worse of the severity of dependence.
Visual analogue scale | 20 months
  The highest score in the whole questionnaire is 10 point, and the lowest score is 0 points. The higher the score, the more serious of the pain.
Clinical Opiate Withdrawal Scale | 20 months
  The highest score in the whole questionnaire is 55 point, and the lowest score is 0 points. The higher the score, the more serious of the Withdrawal symptom.
Beck Depression Inventory | 20 months
  The highest score in the whole questionnaire is 63 point, and the lowest score is 0 points. The higher the score, the more serious of depression.
Beck Anxiety Inventory | 20 months
  The highest score in the whole questionnaire is 63 point, and the lowest score is 0 points. The higher the score, the more serious of anxiety.
The Short Form (36) Health Survey | 20 months
  The highest score in the whole questionnaire is 100 point, and the lowest score is 0 points. The lower the score, the better quality of life.
Craving Scale | 20 months
  The highest score in the whole questionnaire is 108 point, and the lowest score is 0 points. The higher the score, the more serious of craving behavior.

CONTACTS AND LOCATIONS:
Overall Officials: YU Kai-Chiang, Principal Investigator — Chinese Medicine Center Medical Office
Locations (1):
- Department of Chinese Medicine, Taipei City Hospital, Linsen, Chinese Medicine, and Kunming Branch, Taipei, Taiwan, Taipei County, Taipei, Taiwan